CLINICAL TRIAL: NCT01455714
Title: Finding Early Predictors of Myocardial Dysfunction in Patients With Hypertension
Acronym: dysh
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Agata Bielecka-Dabrowa, MD, PhD, Department of Hypertension, MD, PhD, FESC, Principal Investigator, Department of Hypertension, Medical University of Lodz
Other Study IDs: RNN/446/10/KB
Record Dates: First submitted 2011-09-21; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Hypertension
Keywords: hypertenion; exertional dyspnoea; heart failure; biomarkers
MeSH Terms: conditions — Hypertension; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A, B, C: Group A- 40 patients without symptoms of heart failure Group B- 40 patients with exertional dyspnoea Group C - 40 patients with overt heart failure

SUMMARY:
Finding early predictors of myocardial in patients with hypertension

1. Scientific objective The study objective is to clarify the grounds of heart exertional dyspnoea stenocardial pain in patients with well-controlled stage I or II hypertension according to ESH (European Society of Hypertension), without changes in epicardial coronary arteries in coronary angiography and normal resting echocardiography result, and to assess of potential early markers of heart hypertrophy and failure in patients with hypertension.

   Characteristics of the final result The study is to allow for identification of patients with hypertension, in whom an early introduction of pharmacological treatment of heart failure should be considered. Evaluation in the detection of asymptomatic myocardial dysfunction will include potential heart failure markers such as: cardiotrophin 1, cystatin C, serum syndecan-4, collagen III N-terminal propetide [PIIINP], MMP-2, MMP-7, MMP-8, MMP-9 and NT-proBNP, modern echocardiography methods and magnetic resonance imaging in order to increase the effectiveness of prevention, diagnosis and treatment optimalization.
2. Project significance Prognosis in heart failure is very serious. It is similar or worse than in advanced cancer. These data indicate an extreme importance of the optimal early causal treatment of hypertension and symptomatic treatment of heart failure early stage in order to prevent the development advanced form of the disease, which has bad prognosis. In clinical practice, patients with well-controlled hypertension often report exercise limitation, exertional dyspnea and/or stenocardial pain which is not reflected in a standard resting echocardiography (normal result), without coronary artery disease data in electrocardiographic stress test and without change in epicardial coronary vessels in coronary angiography. The study is designed to establish the panel of diagnostic tests in patients with hypertension and exertional dyspnoea only, which will allow for early detection of abnormalities (before symptoms occur) and the start of the optimal treatment for these patients. Unfortunately, still too small percentage of patients receives full pharmacotherapy, hence the authors of the latest guidelines of procedure in heart failure and hypertension put great emphasis on this aspect. Optimal management may prevent the progression of these patients in stage C heart failure, and thus bring tangible benefits not only the patients themselves but also, by reducing the number of costly hospitalizations, significantly reduce health care costs. The number of hospitalizations for heart failure in Poland is estimated at 100 000 per year, and hospitalization costs exceed 70% of the total costs associated with the treatment of heart failure. The issue of exertional dyspnoea and overt heart failure in patients with hypertension and normal results of resting echocardiography is a new problem, both in Poland and in the world.

So far, there are no treatment recommendations for this group of patients. Material and study plan 120 persons (age 40-60 years old) will be included in the study, patients with stage I or II primary hypertension according to the European Society of Hypertension: Group A- 40 patients without symptoms of heart failure Group B- 40 patients with exertional dyspnoea Group C - 40 patients with overt heart failure

In group B (patients with exertional dyspnea/stenocardia) we will include only patients who have undergone contrast coronary angiography without any identified changes in the epicardial coronary arteries, which will facilitate answering the presented purpose of research. Patients in groups A and B with normal resting echocardiography and treated with a maximum of 2 antihypertensive drugs (an ACE inhibitor or a sartan as therapy base), according to the following regimen:

ACEI/ARB + diuretic ACEI/ARB + calcium channel antagonist Group C - treatment in accordance with the standards for heart failure. Each patient will be informed about the objectives of the study and give written consent to participate.

After signing informed consent patients will have performed the following tests:

* Interview and documentation analysis,
* Physical examination,
* Electrocardiogram,
* 24-hour blood pressure monitoring (ABPM),
* 24-hour EKG recording,
* Echocardiography at rest and during submaxinal exercise on a bicycle ergometer,
* Flow-mediated dilatation (FMD),
* Cardiac magnetic resonance imaging,
* Standard labolatory parameters,
* Levels of markers: cystatin C, cardiotrophin-1, metaloproteinases: MMP-2, MMP-7, MMP-8, MMP-9, Procollagen III N-Terminal Propeptide (PIIINP), Syndecan 4 (SDC4) and NT-proBNP Each patient will be informed about the objectives of the study and give written consent to participate.

DETAILED DESCRIPTION:
The concept and plan of study

1. The attempt to clarify the grounds of heart exertional dyspnoea stenocardial pain in patients with well-controlled stage I or II hypertension according to ESH (European Society of Hypertension), without changes in epicardial coronary arteries in coronary angiography and normal resting echocardiography.
2. MRI evaluation of coronary microcirculation and endothelial function assessed by flow-dependent vasodilation in hypertensive patients with and without heart failure symptoms.
3. Comparison of modern echocardiographic methods and magnetic resonance imaging in the diagnosis of hypertensive patients with and without overt heart failure.
4. Cystatin C as a new marker of organ damage in patients with hypertension and comparison of cystatin C with GFR assessed by MDRD and Cockcroft-Gault creatinine clearance on as renal function assessment indicators in patients with hypertension.
5. Evaluation of new markers - cardiotrophin 1 and cystatin C, serum syndecan-4, collagen III N-terminal propetide [PIIINP], MMP-2, MMP-7,MMP-8, MMP-9 and NT-proBNP in the early diagnosis of heart failure.
6. Potential markers of heart failure, modern echocardiography methods and magnetic resonance imaging in the detection of asymptomatic myocardial dysfunction in order to increase the effectiveness of prevention and treatment.
7. Searching for the relationship between the type of hypertension (dipper or non-dipper) and the development of heart failure symptoms, and whether there are differences between the echocardiographic images of these patients?
8. Selection of patients with hypertension, in whom an early introduction of pharmacological treatment of heart failure should be considered.
9. The study will also help answer the following questions: (a) Which parameters best assess the overall cardiovascular risk? and (b) When the treatment of heart failure in patients with hypertension should start.

The measurable effect of this research besides cognitive is to the possibility of reducing the proportion of patients who come to overt heart failure connected with hypertension through the optimization of preventive, diagnostic methods and to determine the optimum treatment in these patients.

ELIGIBILITY:
Inclusion Criteria:

* 120 persons (age 40-60 years old) will be included in the study, patients with stage I or II primary hypertension according to the European Society of Hypertension

Exclusion Criteria:

Following patients will be excluded from the study:

* with coronary artery disease or a history of coronary artery disease
* with unstable hypertension
* with a positive stress test
* with NYHA class III-IV heart failure
* after percutaneous or surgical revascularization
* with diabetes
* with GFR < 60
* with hyperthyroidism and hypothyroidism
* active smokers
* with an implanted pacemaker
* with hip, knee endoprosthesis
* with claustrophobia
* with obesity level II and III
* with ECG-arrhythmia
* pregnant and lactating
* with congenital heart disease
* with hemodynamically significant acquired heart defects
* with cardiomyopathies
* with cancer
* with anemia
* abusing alcohol or drugs
* with chronic inflammatory and other diseases
* or who have not given their informed consent to participate in the study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 120 persons (age 40-60 years old) will be included in the study, patients with stage I or II primary hypertension according to the European Society of Hypertension
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Changes in levels of biomarkers | two years
  Levels of markers: cystatin C, cardiotrophin-1, metaloproteinases: MMP-2, MMP-7, MMP-8, MMP-9, Procollagen III N-Terminal Propeptide (PIIINP), Syndecan 4 (SDC4) and NT-proBNP
echocardiographical parameters | two years
  Echocardiography at rest and during submaxinal exercise on a bicycle ergometer
assessment of perfusion and endothelium function | two years
  * Flow-mediated dilatation (FMD),
  * Cardiac magnetic resonance imaging,

SECONDARY OUTCOMES:
mortality | two years
exertional dyspnoea | two years
heart failure aggravation | two years

CONTACTS AND LOCATIONS:
Overall Officials: Agata Bielecka-Dabrowa, MD, PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Department of Hypertension MU of Lodz, Lodz, Poland